CLINICAL TRIAL: NCT01491568
Title: Pilot Study of Recombinant Human Bone Morphogenetic Protein-2 and Compression Resistant Matrix With the CD HORIZON® Spinal System for Posterolateral Lumbar Fusion in Patients With Symptomatic DDD at Two Adjacent Vertebral Levels
Brief Title: rhBMP-2/CRM/CD HORIZON® Spinal System Pilot Study (2-Level)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04-07
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Degenerative Disc Disease
Keywords: symptomatic degenerative disc disease at two levels
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Investigational (Experimental)
  Interventions: Device: rhBMP-2/CRM/CD HORIZON® Spinal System

INTERVENTIONS:
Device: rhBMP-2/CRM/CD HORIZON® Spinal System — rhBMP-2/CRM with the CD HORIZON® SpinalSystem
  Other Names: Recombinant human bone morphogenetic protein-2

SUMMARY:
The purpose of this study is to evaluate the feasibility of using the investigational implant (rhBMP-2/CRM with the CD HORIZON® Spinal System) as a method of facilitating posterolateral lumbar spinal fusion at two adjacent treatment levels in patients with symptomatic degenerative disc disease.

ELIGIBILITY:
Inclusion Criteria:

1. Has degenerative disc disease at two adjacent lumbar levels as noted by back pain of discogenic origin, with or without leg pain, with degeneration of the disc confirmed by patient history and radiographic studies to include one or more of the following:

   * instability;
   * osteophyte formation;
   * decreased disc height;
   * thickening of ligamentous tissue;
   * disc degeneration or herniation; and/or
   * facet joint degeneration.
2. Has preoperative Oswestry score >= 30.
3. Has no greater than Grade 1 spondylolisthesis utilizing Meyerding's Classification (Meyerding, HW, 1932) at either treatment level.
4. Requires fusion at two adjacent lumbar levels from L1 to S1.
5. Is at least 18 years of age, inclusive, at the time of surgery.
6. Has not responded to non-operative treatment( e.g., bed rest, physical therapy, medications, spinal injections, manipulation, and/or TENS) for a period of 6 months.
7. If a female of child-bearing potential, patient is non-pregnant and non-nursing and agrees to not become pregnant for 1 year following surgery.
8. Is willing and able to comply with the study plan and sign the Patient Informed Consent Form.

Exclusion Criteria:

1. Has primary diagnosis of a spinal disorder other than degenerative disc disease with Grade 1 or less spondylolisthesis at the involved levels.
2. Has had previous spinal fusion surgical procedure(s) at the involved levels.
3. Requires spinal fusion at more than two lumbar levels.
4. Has a condition that requires postoperative medications that interfere with fusion, such as steroids or prolonged use of nonsteroidal anti-inflammatory drugs, excluding routine perioperative nonsteroidal anti-inflammatory drugs. This does not include low dose aspirin for prophylactic anticoagulation.
5. Has been previously diagnosed with osteopenia, osteomalacia, or osteoporosis, or has any of the following that may be associated with a diagnosis of osteoporosis. (If "Yes" to any of the criteria below, a dual x-ray absorptiometry [DEXA] scan will be required to determine eligibility.)

   * Previously diagnosed with osteopenia, osteomalacia, or osteoporosis.
   * Postmenopausal non-black female over 60 years of age who weighs less than 140 pounds.
   * Postmenopausal female who has sustained a nontraumatic hip, spine, or wrist fracture.
   * Male over the age of 70.
   * Male over the age of 60 who has sustained a nontraumatic hip or spine fracture. If the level of bone mineral density (BMD) is a T score of -3.5 or lower( i.e., -3.6, - 3.7, etc.) or a T score of -2.5 or lower( i.e., -2.6,
   * 2.7, etc.) with vertebral crush fracture, then the patient is excluded from the study.
6. Has presence of active malignancy or prior history of malignancy (except for basal cell carcinoma of the skin).
7. Has overt or active bacterial infection, either local or systemic.
8. Has a documented titanium alloy allergy or intolerance.
9. Is mentally incompetent. If questionable, obtain psychiatric consult.
10. Has a Waddell Signs of Inorganic Behavior Score of 3 or greater.
11. Is a prisoner.
12. Is an alcohol and/or drug abuser as defined by currently undergoing treatment for alcohol and/or drug abuse.
13. Has received drugs that may interfere with bone metabolism within two weeks prior to the planned date of spinal fusion surgery( e.g., steroids or methotrexate).
14. Has a history of autoimmune disease.
15. Has a history of exposure to injectable collagen or silicone implants.
16. Has a history of hypersensitivity to protein pharmaceuticals (monoclonal antibodies or gamma globulins) or collagen.
17. Has received treatment with an investigational therapy within 28 days prior to implantation surgery or such treatment is planned during the 16 weeks following rhBMP-2/CRM implantation.
18. Has received any previous exposure to any/all BMPs of either human or animal extraction.
19. Has a history of allergy to bovine products or a history of anaphylaxis.
20. Has history of endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's disease, renal osteodystrophy, Ehlers-Dalons syndrome, or osteogenesis imperfecta).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2005-07; Primary Completion 2009-05 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Overall Success | 24 month
  A patient will be considered an overall success if all of the following conditions are met:
  1. fusion;
  2. pain/disability (Oswestry) improvement;
  3. maintenance or improvement in neurological status;
  4. no serious adverse event classified as "implant associated", or "implant/surgical procedure associated";
  5. no additional surgical procedure classified as a "failure".

SECONDARY OUTCOMES:
General health status (SF-36) | 24 month
Pain status (back pain, leg pain) | 24 month
Patient satisfaction | 24 month
Patient global perceived effect | 24 month